CLINICAL TRIAL: NCT04403685
Title: Safety and Efficacy of Tocilizumab in Moderate to Severe COVID-19 and Increased Inflammatory Markers: a Phase III Randomized Clinical Trial (COVID-19 Coalition Brazil VI) (TOCIBRAS)
Brief Title: Safety and Efficacy of Tocilizumab in Moderate to Severe COVID-19 With Inflammatory Markers
Acronym: TOCIBRAS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Safety
Sponsor: Beneficência Portuguesa de São Paulo (Other)
Collaborators: Hospital do Coracao (Other); Hospital Israelita Albert Einstein (Other); Hospital Sirio-Libanes (Other); Hospital Alemão Oswaldo Cruz (Other); Brazilian Research In Intensive Care Network (Network); Hospital Moinhos de Vento (Other); Brazilian Clinical Research Institute (Other); Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Dr Rozana Mesquita Ciconelli, Head of research team, Beneficência Portuguesa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOCIBRAS
Record Dates: First submitted 2020-05-24; First posted 2020-05-27 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: COVID; SARS Pneumonia; Cytokine Release Syndrome
Keywords: SARS-CoV 2; SARS Pneumonia; Tocilizumab; Cytokine release syndrom; Interleukin-6; Hyperinflammation
MeSH Terms: conditions — Cytokine Release Syndrome | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, superiority, open-label, controlled trial. Randomization 1:1 to best supportive care (BSC) versus Tocilizumab + BSC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tocilizumab (Experimental): Single-dose tocilizumab of 8 mg/kg (maximum dose of 800mg). Best supportive care.
  Interventions: Drug: Tocilizumab
- Control arm (No Intervention): Best supportive care.

INTERVENTIONS:
Drug: Tocilizumab — Single-dose infusion of 8 mg/kg. Maximum dose of 800 mg.
  Other Names: Actemra
  Arms: Tocilizumab

SUMMARY:
The trial evaluates the efficacy and safety of Tocilizumab, which rapidly reduces the inflammation process through inhibition of IL-6 in patients with moderate to severe COVID-19 with increased inflammatory markers. There will be two arms in the trial, one receiving the best supportive care, and the other receiving it plus tocilizumab. Patients will be followed until Day 29 after randomization.

DETAILED DESCRIPTION:
Coalition VI (TOCIBRÁS) is a prospective phase III randomized controlled trial that evaluates the efficacy and safety of Tocilizumab, an antibody anti-IL-6 receptor in patients with moderate to severe COVID-19 with increased inflammatory markers. This is a superiority open-label study with two arms. The control arm receives the best supportive care, and the experimental receives it plus tocilizumab. Randomization is done centrally by REDCap 1:1. Patients will be followed until Day 29 after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Male and females with 18 years and older
* Confirmed diagnosis of SARS-CoV 2 infection
* More than 3 days of symptoms related to COVID-19
* Computed tomography (or Chest X-Ray) with COVID-19 alterations
* Both of the criteria

  1. Need for oxygen supplementation to keep SPO2 > 93% OR need for mechanical ventilation for less than 24 hours before the randomization
  2. At least two of the following inflammatory tests above the cutoff :

     1. D-dimer > 1,000 ng/mL
     2. Reactive C protein > 5 mg/dL
     3. Ferritin > 300 mg/dL
     4. Lactate dehydrogenase > upper level limit

Exclusion Criteria:

* Need for mechanical ventilation for 24 hours or more before the randomization
* Hypersensitivity to tocilizumab
* Patients without therapeutic perspective or in palliative care
* Active non controlled infections
* Other clinical conditions that contraindicate tocilizumab, according to the assistant physician
* Low neutrophils count (< 0.5 x 109/L)
* Low platelets count (< 50 x 109/L)
* Liver disease, cirrhosis or elevated AST or ALT above 5 times the upper level limit
* Renal disease with estimate glomerular filtration below 30 mL/min/1.72 m2 (MDRD or CKD-EPI scores)
* Active diverticulitis
* Breastfeeding women
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Evaluation of clinical status | Day 15 of the trial
  Evaluation of clinical status of patients on day 15 after randomization, defined by the Ordinal Scale of 7 points (score ranges from 1 to 7, with 7 being the worst score)

SECONDARY OUTCOMES:
All-cause mortality | 29 days after the randomization
  All-cause mortality from randomization to day 28
Hospital Mortality | 29 days after the randomization
  Deaths that occur during hospital admission.
Improvement of Sequential Sepsis-related Organ Failure Assessment (SOFA) scale | 29 days after the randomization (evaluations at D8 and D15)
  Improvement of SOFA scale of patients at day 8, 15 and 29 after randomization
Evaluation of clinical status | 29 days after the randomization (evaluations at D8 and D29)
  Evaluation of clinical status of patients on the day 8, 22 and 29 after randomization, defined by the Ordinal Scale of 7 points (score ranges from 1 to 7, with 7 being the worst score)
Ventilator free days | 29 days after the randomization
  Days alive and free from mechanical ventilation since randomization
Time until oxygen support independence | 29 days after the randomization
  Days from randomization to independence of oxygen support
Need of mechanical ventilation support | 29 days after the randomization
  Number of patients that were not at mechanical ventilation at randomization and that required that support.
Days to mechanical ventilation support. | 29 days after the randomization
  Number of days to mechanical ventilation for patients that were not receiving it at randomization.
  For patients that were not in mechanical ventilation at randomization: number of days until that support was required.
Duration of hospitalization | 29 days after the randomization
  Lenght of hospitalization stay in survivors (in days)
Other infections | 29 days after the randomization
  Incidence of other infections (aside from SARS-CoV 2)
Incidence of thromboembolic events | 29 days after the randomization
  Incidence of thromboembolic events in patients with COVID-19
Incidence of adverse events | 29 days after the randomization (specific evaluations at D8, D15 and D29)
  Evaluation of adverse events, as well as serious and unexpected adverse events

OTHER OUTCOMES:
Correlation of inflammatory tests and cytokines with clinical outcomes | 29 days after the randomization
  Correlation of inflammatory tests and cytokines with clinical outcomes: clinical status (ordinal scale), time to oxygen support independence, ventilator free days, need of mechanical ventilation and mortality
Exploratory evaluation of laboratory exams during hospitalization | 29 days after the randomization
  Evaluation the kinetics of hemostasia exams, inflammatory tests, cytokines, flow cytometry of blood cells, CBC, renal and liver exams
Evaluation of viral clearance of SARS-CoV2 | Day 8 and 15 after randomization
  Evaluation of viral clearance of SARS-CoV2 using RT-PCR analysis of nasopharyngeal swab

CONTACTS AND LOCATIONS:
Overall Officials: Viviane C Veiga, MD, Principal Investigator — Beneficência Portuguesa de Sao Paulo
Locations (7):
- Brazil (7):
  - HCOR -Hospital do Coracao, São Paulo, São Paulo
  - UNIFESP, São Paulo, São Paulo
  - HAOC - Hospital Alemao Oswaldo Cruz, São Paulo
  - Beneficência Portuguesa de Sao Paulo, São Paulo
  - HAOC - Hospital Alemao Oswaldo Cruz - unidade Vergueiro, São Paulo
  - HIAE - Hospital Israelita Albert Einstein, São Paulo
  - HSL - Hospital Sírio Libanês, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Veiga VC, Prats JAGG, Farias DLC, Rosa RG, Dourado LK, Zampieri FG, Machado FR, Lopes RD, Berwanger O, Azevedo LCP, Avezum A, Lisboa TC, Rojas SSO, Coelho JC, Leite RT, Carvalho JC, Andrade LEC, Sandes AF, Pintao MCT, Castro CG Jr, Santos SV, de Almeida TML, Costa AN, Gebara OCE, de Freitas FGR, Pacheco ES, Machado DJB, Martin J, Conceicao FG, Siqueira SRR, Damiani LP, Ishihara LM, Schneider D, de Souza D, Cavalcanti AB, Scheinberg P; Coalition covid-19 Brazil VI Investigators. Effect of tocilizumab on clinical outcomes at 15 days in patients with severe or critical coronavirus disease 2019: randomised controlled trial. BMJ. 2021 Jan 20;372:n84. doi: 10.1136/bmj.n84. PMID 33472855